CLINICAL TRIAL: NCT02768675
Title: Intra-Operative Assessment of the Intellirod LOADPRO Disposable Spinal Rod Strain Sensor for Use During Kyphotic Corrective Surgery
Brief Title: Intra-operative Assessment of the Intellirod LOADPRO Spinal Rod Strain Sensor for Use During Kyphotic Corrective Surgery
Acronym: LOADPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intellirod Spine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LOADPRO EX-0029
Record Dates: First submitted 2016-05-05; First posted 2016-05-11 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Kyphosis; Spinal Fractures
Keywords: Kyphotic; Corrective Surgery; Spinal fractures
MeSH Terms: conditions — Kyphosis; Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LOADPRO arm (Experimental): Participants will temporarily receive a LOADPRO device affixed to kyphotic corrective rods. The device will not be implanted and will be removed prior to surgery closure.
  Interventions: Device: LOADPRO

INTERVENTIONS:
Device: LOADPRO — The Intellirod LOADPRO sensor is a single-use, disposable instrument for the intra-operative measurement of posterior instrumented, spine rod strain.

SUMMARY:
The LOADPRO Study is an intra-operative, non-significant risk (NSR) case series feasibility assessment of the Intellirod LOADPRO™ System measuring spinal rod strain in long spinal kyphotic corrective constructs.

DETAILED DESCRIPTION:
The Intellirod LOADPRO™ sensor is an intra-operative titanium and ceramic, single use, disposable, strain sensing device, which includes hermetically sealed, micro electromechanical systems (MEMS) and radio-frequency identification (RFID) technology to enable measurement of intra-operative rod strain values. The transponder attaches to any commercially available 5.5mm diameter CoCr or Ti Alloy rod commonly used for posterior pedicle fixation systems. The transponder is used only to acquire rod strain values and a unique device identification code, which is obtained by a hand-held reader, providing real-time, objective measurement of the mechanical rod strain.

This non-significant risk case series is intended to assess the effectiveness of the Intellirod LOADPRO™ sensor methodology and the intra-operative measurement of spinal rod strain. The LOADPRO™ sensors will be removed from the spinal rods after obtaining load measurements.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age
* presenting with a confirmed diagnosis of kyphosis with deformity greater than 70 degrees requiring large segmental correction involving a minimum of six (6) levels
* failure of conservative therapy requiring surgical correction of sagittal imbalance
* sagittal imbalance due to loss of lumbar lordosis, and/or segmental kyphosis
* participated in the informed consent process and has signed an Institutional Review Board approved informed consent

Exclusion Criteria:

* women who are pregnant
* evidence of active (systemic or local) infection at time of surgery
* prisoner or transient
* history of known narcotic abuse
* psychological disturbance past or present that could impair the consent process or ability to complete subject self-report questionnaires
* ASA > 3
* osteoporosis diagnosed on DEXA defined as a T-score ≥ -2.0
* Unable or unwilling to provide a full informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Bilateral Rod Strain Readings | Intra-operative
  In this research study, the LOADPRO device will be used solely to monitor and record rod strain readings. The device is not intended, and won't be used, to control or make any rod adjustments by the operative surgeon. In order to provide assurance that the readings cannot be used to make adjustments intra-operatively, the surgeon investigators will be blinded to the rod strain measurement readings.

OTHER OUTCOMES:
Back and bilateral leg pain | up to 1 year post-procedure
  (0 to 10) rating scale
Patient Questionnaire | up to 1 year post-procedure
  Scoliosis Research Society 22-r

CONTACTS AND LOCATIONS:
Overall Officials: Richard N Navarro, Study Director — Intellirod Spine
Locations (2):
- United States (2):
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - OhioHealth Neurological Physicians, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No